CLINICAL TRIAL: NCT00925665
Title: Intubation of Patients With Odontogenic Abcesses Glidescope vs. Macintosh Technique
Brief Title: Intubation of Patients With Odontogenic Abcesses
Status: Completed | Type: Observational
Sponsor: Kliniken Essen-Mitte (Other)
Responsible Party: Prof.Dr. Harald Groeben, Kliniken Essen-Mitte
Other Study IDs: OdoAbGldscp
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2009-06

CONDITIONS: Odontogenic Abscess
Keywords: Intubation; Glidescope; Macintosh; Abscess; Difficult intubations in patients with odontogenic abscesses
MeSH Terms: conditions — Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glidescope: Patients intubated with the Glidescope technique
  Interventions: Device: Glidescope
- Macintosh: Patients intubated via the conventional direct laryngoscopy with a Macintosh laryngoscope
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: Glidescope — Patients are to be intubated using the Glidescope technique
  Groups: Glidescope
Device: Macintosh laryngoscope — Patients are to be intubated using direct laryngoscopy with a Macintosh laryngoscope
  Groups: Macintosh

SUMMARY:
This study is a comparison of two techniques for endotracheal intubation (Glidescope versus Macintosh) in patients with odontogenic abscesses.

DETAILED DESCRIPTION:
Patients with odontogenic abcesses have to be treated by surgical drainage of the abscess under general intubation with endotracheal intubation. Because of a limited mouth opening and swelling within the oral cavity, intubation can be difficult and sometimes impossible with conventional direct laryngoscopy. Therefore, alternative techniques are desirable. We want to compare the success rate of intubation in these patients using the Glidescope technique vs. conventional Macintosh technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to have an abscess which has to be treated surgically.
* Mouth opening (Inter-incisor gap) has to be less than 3.5 cm and more than 1.4 cm.

Exclusion Criteria:

* Age under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We want to study patients, who present with a odontogenic abscess for surgical treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Success rate of endotracheal intubation | 18 months

SECONDARY OUTCOMES:
Time for intubation | 18 months
View of the laryngeal entrance (according to the classification of Cormack and Lehane) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Harald Groeben, M.D., Principal Investigator — Kliniken Essen-Mitte
Locations (1):
- Kliniken Essen-Mitte, Essen, Germany

REFERENCES:
- [Background] Arne J, Descoins P, Fusciardi J, Ingrand P, Ferrier B, Boudigues D, Aries J. Preoperative assessment for difficult intubation in general and ENT surgery: predictive value of a clinical multivariate risk index. Br J Anaesth. 1998 Feb;80(2):140-6. doi: 10.1093/bja/80.2.140. PMID 9602574